CLINICAL TRIAL: NCT04916483
Title: Exploring the Effectiveness of Group Cognitive Stimulation Therapy on Cognitive Function, Depressive Symptoms, Social Function and Quality of Life in People With Schizophrenia: A Randomized Controlled Trial
Brief Title: Exploring the Effectiveness of Group Cognitive Stimulation Therapy in People With Schizophrenia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Chiu-Yueh Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB1081209-04
Record Dates: First submitted 2020-04-09; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Cognitive Therapy
Keywords: cognitive stimulation therapy; depressive symptoms; schizophrenia; social function; quality of life
MeSH Terms: conditions — Depression; Schizophrenia; Social Adjustment

STUDY DESIGN:
Intervention Model Description: Participants were divided into experimental group and control group through block randomization
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The questionnaire is distributed and applied by another researcher (non-investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exploring the effectiveness of GCST in people with schizophrenia. (Experimental): The experimental group will receive a total of 14 sessions, twice a week group cognitive stimulation therapy for 7 weeks.
  Interventions: Other: group cognitive stimulation therapy; Other: usual care
- Control group (No Intervention): The control group maintains the usual care.

INTERVENTIONS:
Other: group cognitive stimulation therapy — The experimental group will receive totally 7 weeks,14 sessions, twice a week, and 60 minute group cognitive stimulation therapy (GCST).
  Other Names: GCST
  Arms: Exploring the effectiveness of GCST in people with schizophrenia.
Other: usual care — The control group maintains the unit routine treatment.
  Arms: Exploring the effectiveness of GCST in people with schizophrenia.

SUMMARY:
Background: Cognitive dysfunction is the core defect of schizophrenia, which seriously affects the emotional, social functions and quality of life in people with schizophrenia.

Objective: The purpose of this study is to explore the efficacy of group cognitive stimulation therapy in cognitive function, depressive symptoms, social function, and quality of life in people with Schizophrenia.

Research method:This study used a single-blind randomized controlled trial design. Participants's Montreal Cognitive Assessment Scale (MoCA) score between 10-25 points are include. Chronic rehabilitation wards were randomly assigned to the experimental group and the conventional treatment group using blocking. The experimental group (EG) (n = 45) is receive 7 weeks, twice a week, 60 minutes each time of group cognitive stimulation therapy(GCST), the control group (CG) (n = 45) maintain usual care.

Expected results: GCST can improve cognitive function, depressive symptoms, social function and quality of life in people with schizophrenia.

DETAILED DESCRIPTION:
Background: Cognitive dysfunction is the core defect of schizophrenia, which seriously affects the emotional and social functions of patients. Group cognitive stimulation therapy has been supported by research abroad to improve cognition and mood. Domestically, this group of people with schizophrenia will also face the above symptoms. Therefore, non-pharmacological therapy is among mental health personnel It is worth paying attention to and developing in the process of providing medical services.

Objective: The purpose of this study explores the efficacy of group cognitive stimulation therapy in cognitive function, depressive symptoms, social function and quality of life in people with Schizophrenia.

Research method: This study used a single-blind randomized controlled trial design to reduce it to people with schizophrenia.This study used a single-blind randomized controlled trial design. Participants's Montreal Cognitive Assessment Scale (MoCA) score between 10-25 points are include. Chronic rehabilitation wards were randomly assigned to the EG and the CG using blocking. The EG receive 7 weeks, twice a week, 60 minutes each time of GCST, the CG maintain usual care. Both groups use the Montreal Cognitive Assessment Scale (MoCA), the Taiwanese Version of Frontal Assessment Battery (TFAB), the Beck Depression Inventory II (Beck Depression Inventory II, BDI-II), and Social Function Scales-Taiwanese version(SFST) and WHOQOL-BREF is use as an evaluation tool to measure the results at the baseline, T1 (7th weeks) and T2 (20th weeks). The research results were filed and statistically analyzed with IBM SPSS 20.0 software package. Descriptive statistics were used for general demographic variables and primary , secondary outcome: mean, SD, range, percentage. The difference between the two groups of benchmark values was analyzed with t-test or χ2, independent-t test, pair-t, and GEE.

Expected results: GCST can improve cognitive function, depressive symptoms, social function and quality of life in people with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. People who according the DSM-5 diagnosis of schizophrenia spectrum and have been sick for more than two years.
2. Age between 20 and 65 years old.
3. There are currently rules for receiving antipsychotics treatment.
4. Regardless of whether you take antidepressants or not.
5. Can communicate clearly in Mandarin and Taiwanese.
6. Those with a score of 10-25 on the Montreal Cognitive Assessment Scale (MoCA).
7. Those who are willing to participate in this study and complete the subject consent form.

Exclusion Criteria:

1. According to DSM-5 criteria, suspected bipolar disorder, anxiety disorder, obsessive- compulsive disorder, cognitive impairment, substance use disorders, and other unthinking disorders are exclusion.
2. Have been in or out of the acute ward within three months and currently have suicidal attempts or violence.
3. Those who are receiving individual or group cognitive behavior therapy.
4. People with intellectual disabilities.
5. Those who are unable to conduct research due to visual or hearing impairment.
6. People who are accepting other clinical trials.
7. Those who have no intention to participate in this study or are unable to complete the subject's consent form.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment, MoCA | baseline
  Cognitive function test
Taiwanese Version of Frontal Assessment Battery, TFAB | baseline
  Cognitive function test
Wechsler Memory Scale-Third Edition, WMS-III | baseline
  Cognitive function test

SECONDARY OUTCOMES:
Beck Depression Inventory II, BDI-II | baseline
  Depressive symptoms test
Social Function Scales-Taiwanese version, SFST | baseline
  Social Function test
WHOQOL-BREF | baseline
  quality of life test

OTHER OUTCOMES:
Montreal Cognitive Assessment, MoCA | 7th weeks
  Cognitive function test
Taiwanese Version of Frontal Assessment Battery, TFAB | 7th weeks
  Cognitive function test
Wechsler Memory Scale-Third Edition, WMS-III | 7th weeks
  Cognitive function test
Beck Depression Inventory II, BDI-II | 7th weeks
  Depressive symptoms test
Social Function Scales-Taiwanese version, SFST | 7th weeks
  Social Function test
WHOQOL-BREF | 7th weeks
  quality of life test
Montreal Cognitive Assessment, MoCA | 20th week
  Cognitive function test
Taiwanese Version of Frontal Assessment Battery, TFAB | 20th week
  Cognitive function test
Wechsler Memory Scale-Third Edition, WMS-III | 20th week
  Wechsler Memory Scale-Third Edition, WMS-III
Beck Depression Inventory II, BDI-II | 20th week
  Depressive symptoms test
Social Function Scales-Taiwanese version, SFST | 20th week
  Social Function test
WHOQOL-BREF | 20th week
  quality of life test

CONTACTS AND LOCATIONS:
Overall Officials: Chiu-Yueh Yang, PhD, Principal Investigator — National Yang-Ming Jiaotong University
Locations (1):
- National Yang-Ming Jiaotong University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No